CLINICAL TRIAL: NCT04698291
Title: Identifying the Effect of Genetic Variants on Specialized Pro-resolving Mediators and Their Association With Chronic Inflammatory Conditions
Brief Title: Genetic Variants and Regulation of Specialized Pro-resolving Mediator
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 291815
Record Dates: First submitted 2020-12-18; First posted 2021-01-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Inflammatory Disease; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Blood Donation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: This research aims to recruit only adult volunteers that have taken part of the Gene & Health program. We will focus on two groups: individuals presenting the polymorphisms of interest and individuals without the genetic variants in the genes of interest, which will be used as matched controls. Eligible individuals will consent to donate blood samples for this study, in addition to consent access to their medical and health records.
  Interventions: Procedure: Blood Donation
- Cases: This research aims to recruit only adult volunteers that have taken part of the Gene & Health program. We will focus on two groups: individuals presenting the polymorphisms of interest and individuals without the genetic variants in the genes of interest, which will be used as matched controls. Eligible individuals will consent to donate blood samples for this study, in addition to consent access to their medical and health records.
  Interventions: Procedure: Blood Donation

INTERVENTIONS:
Procedure: Blood Donation — The blood donation will take place at the Gene & Health clinical assessment centre facilities. A trained member from Gene & Health program will be responsible for taking the blood samples.

SUMMARY:
Inflammation is the way that the body reacts against infection, injury or illness. An uncontrolled inflammatory response can lead to the development of inflammatory diseases, such as rheumatoid arthritis and cardiovascular conditions. Recent studies have shown that inflammation is a regulated process coordinated by a group of molecules known as specialized pro-resolving mediator (SPM). These molecules are produced by enzymes via the enzymatic conversion of essential fatty acids; whereas their biological actions are mediated by proteins expressed on the surface of cells known as receptors.

Given the central role that pro-resolving mediators play in regulating the immune response, the aim of this study is to investigate whether there are genetic variants (mutations) in genes encoding for enzymes and receptors involved in the biology of these molecules and to determine how these mutations affect SPM's activity or function.

Findings made as part of these studies will help shed light into mechanism influencing disease onset and/or progression and potentially enhance the discovery of new and more effective treatments.

DETAILED DESCRIPTION:
This study aims to identify polymorphisms in SPM-related genes in a South Asian population and assess whether these lead to alterations in the functions of enzymes and proteins encoded by these genes. This information will then be used to identify those SNP (Single nucleotide polymorphism) that lead to loss of function. We will then evaluate whether these SNP are linked with altered white blood cell function and increased incidence of chronic inflammatory disorders by assessing data from the Gene & Health program and other databases such as UK Biobank. We expect that this approach will provide new insights into molecular mechanisms and the identification of new mediators/enzyme/receptors families that are dysregulated in inflammatory conditions.

To achieve this aim, we will identify volunteers from the Gene & Health program. The Gene & Health program has sequenced around 40,000 volunteers and identified around 500 gene variants that are predicted to lead to complete loss of gene function; among these SNP, 68 are presented in enzymes and receptors related with SPM including ALOX15, GPR18 and FPR2/ALX. As part of their recruitment to Gene & Health program, participants have consented to be contacted about future research studies such as this.

In order to study the differences in the lipid mediator profiles between the groups, we will use peripheral blood obtained from consented Gene & Health individuals that present the SNP of interest (cases) and individuals without the mutation (controls). For the lipid mediator profiling a liquid chromatography in tandem mass spectrometry strategy (LC-MS/MS) will be used. Cell biology assays (phagocytosis, platelet activation, etc.) will be conducted using peripheral blood phagocytes cells. In addition, volunteers will be consented for access to their centralised health records so we can identify associations between different polymorphisms and the development of inflammatory conditions through a candidate-gene association study.

The risks of this study to participants are low and relate to the sharing of confidential data and blood sample donation. Access to confidential clinical information with person-identifiable data will be restricted to the Chief Investigator and Principal Investigator, who are aware of their responsibilities under the Data Protection Act 2018 and all the obligations related to data management enforced by Gene & Health program. As for the blood donation, we believe that there is minimal risk to participants as they will only be asked to donate up to 60 ml of blood per sitting and donors will not be recalled more than 3 separate occasions.

ELIGIBILITY:
Inclusion Criteria:

* Current volunteer of the Genes & Health program with (test) or without (control) relevant genetic mutations. Genes & Health is a huge long-term study of 100,000 people of Bangladeshi and Pakistani origin focuses to link genes with health records and to study disease and treatments. When a volunteer participates in this program, they agree to the possibility to be invited for further studies. Gene & Health program invites volunteers to take part in two regions of the UK: East London and Bradford.

Exclusion Criteria:

1. Volunteer that has not had their genome sequenced after taking part in Stage 1 of Genes & Health program.
2. Volunteer with significant genetically inherited conditions.
3. Any abnormality or pre-existing disease which, in the opinion of the investigator, might either expose the subject to risk, or influence the validity of the results.
4. Volunteer that went under surgery and are recovering.
5. Participation in a clinical study of a new chemical entity, biological product or a prescription medicine, or loss of more than 400 mL blood, within the previous 3 months.
6. Presence or history of drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Genes & Health is a huge long-term study of 100,000 people of Bangladeshi and Pakistani origin focuses to link genes with health records and to study disease and treatments. We will be focused on those volunteers with specific mutations in Specialized pro-resolving mediators enzymes and receptors.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2027-10-05 (Estimated); Study Completion 2027-12-08 (Estimated)

PRIMARY OUTCOMES:
Lipid Mediator Profiling | Inmediately after blood sample collection.
  The blood samples will be used to get the lipid mediator profiling (specialized pro-resolving mediators abundance in blood) using a liquid chromatography in tandem mass spectrometry strategy).

SECONDARY OUTCOMES:
Phagocytosis | Up to 6 month after blood sample collection.
  Phagocytosis will be assayed in vitro by measuring the engulfment of Escherichia coli by T cells and Macrophage. The extent of phagocytosis will be assessed using flow cytometry.
Platelet activation | Up to 6 month after blood sample collection.
  Adhesion molecule expression as well as platelet-leukocyte aggregates will be assessed using flow cytometry.
Peripheral blood T-cell assay | Up to 6 month after blood sample collection.
  T-cell activity will be assessed using cytokine expression as well as the expression of activation markers by flow cytometry.
Peripheral blood SPM pathways | Up to 6 month after blood sample collection.
  Enzyme and receptor expression associated with specialized pro resolving mediators will be assessed using flow cytometry.

OTHER OUTCOMES:
Genetic variants associations | 6 months after patient recruitment.
  In addition, volunteers will consent for access to their centralised health records so we can identify associations between different mutations and the development of inflammatory conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jesmond Dalli, Professor, Study Director — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Any results arising from this study will be kept to support future research projects. The information will only be released to recognised researchers whose project has been approved by ethics and medical research committees in the UK. The researchers may be given access to some information about the volunteers health, but will not be given any personal information that can be used to identify them.

REFERENCES:
- See also: Gene & Health program information — http://www.genesandhealth.org/